CLINICAL TRIAL: NCT03641781
Title: Comparison Of Isometric And Isokinetic Strength Training Effects On Physical Performance In Athletes With Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Hafiz Muhammad Manan Haider Khan, Principal investigator, Isra University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIRS-IUISB/PHD/006
Record Dates: First submitted 2018-08-15; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Knee Injuries
Keywords: Isokinetic, Isometric, Agility; Athletic Single Leg Stability,; Vertical Jump Biodex, Knee Pain
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Intervention Model Description: Athletes were randomly assigned into two groups: Isometric (ISOM) and Isokinetic (ISOK). A coin was flipped at start of data collection for the first patient to be assigned odd number and included in isometric group. Later on odd and even numbered patients were included in specific group. Additionally, data was collected from healthy athletes doing their training at Pakistan Sports Board, called healthy control group. Due to ethical constraints knee pain athletes were not included as control subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isometric strength training group (Active Comparator): Knee pain athletes were assessed by The International Knee Documentation Committee (IKDC) 2000 Subjective Knee evaluation form and were assigned into ISOM group. ISOM group participants were involved in isometric strengthTraining at angle of 30°,45°,60° of knee flexion for 5 maximum contraction for both hamstring and quadriceps. 10 sessions were given on alternate day basis by using Biodex Isokinetic system.
  Interventions: Other: isometric strength training and isokinetic strength training
- Isokinetic strength training group (Active Comparator): Knee pain athletes were assessed by The International Knee Documentation Committee (IKDC) 2000 Subjective Knee evaluation form and were assigned into ISOK group isokinetic training group randomly. ISOk group participants were involved in Training at speed of 30 deg/sec, 90deg/sec, 150/deg/sec 210deg/sec, 270deg/sec 5 repetition for both hamstring and quadriceps. 10 sessions were given on alternate day basis by using Biodex Isokinetic system.
  Interventions: Other: isometric strength training and isokinetic strength training
- Healthy control group (No Intervention): Data for outcome parameters including Peak torque average peak torque average power agonist antagonist ratio by using biodex isokinetic system for both by isometric contraction method and isokinetic method. For performance test were recorded for healthy control of same age group to compare the training effect with healthy control values.

INTERVENTIONS:
Other: isometric strength training and isokinetic strength training — Isokinetic strength program included strength training at 5 different velocities from slow to fast. Participants were trained on speed of 30°/sec, 90°/sec, 150°/sec, 210°/sec and 270°/sec. Flexion and extension movements were completed with 5 repetitions at each speed.
  Participants of isometric strength training group performed isometric contractions at 30°, 45° and 60° of knee flexion with five repetitions at each angle for both hamstring and quadriceps.
  Arms: Isokinetic strength training group; Isometric strength training group

SUMMARY:
Frequent sports events causing more injuries in athletes causing decline in their performance. Injuries around knee joint are common. Strength training of hamstring and quadriceps are effective tool in rehabilitation. The multi-speeds and multi-angles strength training plans were used to see the effects on symptoms and performance in athletes.

DETAILED DESCRIPTION:
A total of 69 athletes with knee pain were recruited and randomly divided into two groups. 50 athletes completed the training programs, 25 in each group. Data was also collected from healthy athletes for normative values. International Knee Documentation Committee subjective knee evaluation form was used to report the athlete's knee condition and severity of symptoms including pain. Biodex isokinetic system was used for isokinetic and isometric strength trainings and kinetic data collection. Physical performance of an athlete was assessed by components of fitness through two commonly used tests: Illinois agility run test and vertical jump test. The athletic single leg stability test was used to assess the stability of athletes on Biodex Balance System.

ELIGIBILITY:
Inclusion Criteria:

* The adult athletes between ages 18 to 35 years.
* Athletes with unilateral knee pain.
* Both male and female.

Exclusion Criteria:

* Athletes with bilateral knee pain and any deformity around knee were excluded from this study.
* Any other joint involvement of lower limb while assessment were also excluded from study.
* Athletes with recent history of surgeries for fractures or ligamentous reconstruction were excluded from this study.
* Patients who were medically unstable.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
change in Agility Run Test time | change from baseline through completion an average of 3 weeks
  The agility run test was conducted by placing cones at the non-slippery surface. The time to complete the test was recorded by using stop watch. A 10 Meter distance in figure of 8 was made on ground with help of cones. Time taken to complete was recorded in seconds.
change in Vertical Jump test height | change from baseline through completion an average of 3 weeks
  Vertical jump test was conducted by using the measuring tape placed on wall. Athletes were standing along the wall and the standing height, the highest level of finger touching the wall was recorded initially. Athlete then jumped vertically and marked on the wall and performed three repetitions. The greatest difference between initial standing height and after jump height was recorded as score of vertical jump.
change in Athletic single leg stability test | change from baseline through completion an average of 3 weeks
  The athletic single leg stability test was used to assess the stability of athlete conducted by using Biodex Balance System SD (Biodex Medical Systems, Inc. NY, USA). Athletes were standing on involved leg and platform setting was at level 4. Athletes performed 3 repetitions of 20 seconds each with 10 seconds rest between the repetitions to complete the test. Overall stability index, anterior posterior index, and medial lateral index were recorded.

SECONDARY OUTCOMES:
change in Peak Torque value (FT-LB) | change from baseline through completion an average of 3 weeks
  Highest muscular force output at any moment during a repetition. Peak torque indicates the muscle's maximum strength capability. This is also equivalent to a 1-repetition maximum (RM) isotonic strength test.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR